CLINICAL TRIAL: NCT05246722
Title: Registry Study of Pharmacotherapy and Clinical Outcomes in Elderly Patients With Coronary Heart Disease
Brief Title: Registry Study of Pharmacotherapy and Clinical Outcomes in Elderly Patients With Coronary Heart Disease (PHARM-ageing)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Lin Yang, Director of pharmacy department of Beijing Anzhen Hospital, Beijing Anzhen Hospital
Other Study IDs: ANZHEN HOSPITOL-LY-03
Record Dates: First submitted 2022-01-13; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Elderly Patients; Coronary Heart Disease; Drug Therapy; Clinical Outcomes
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A registry study on drug therapy and clinical outcomes in elderly patients with coronary heart disease

ELIGIBILITY:
Inclusion Criteria:

* Informed consent has been signed
* Patients diagnosed in our hospital with coronary heart disease
* Age ≥65 years

Exclusion Criteria:

* Severe lack of important information such as history of previous medication, history of previous disease, history of surgery.
* Mental disorders, or inability to communicate effectively with researchers, or failure to comply with research protocols.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (≥65 years) with coronary heart disease who discharged at Beijing Anzhen Hospital from January 1, 2019.Those who fill the inclusion criteria at screening will be invited for the registry study.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
main adverse cardiovascular and cerebrovascular events (MACCE) | up to 3 years
  MACCE will be defined as all-cause death, non-fatal stroke, non-fatal myocardial infarction (MI), and ischemic-driven revascularization

SECONDARY OUTCOMES:
Adverse drug reaction | up to 3 years
  Adverse drug reaction will be defined as any adverse reactions in the patients